CLINICAL TRIAL: NCT01146327
Title: A Phase 1, Parallel, Randomized Trial To Assess The Effect Of Time Of Dosing On The Pharmacodynamics, Pharmacokinetics, Safety And Tolerability Of Multiple Oral Doses Of PF-04620110 In Otherwise Healthy Overweight Or Obese Adult Subjects
Brief Title: A Multiple Dose Study Of PF-04620110 In Healthy Overweight Or Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B0961010
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Healthy
Keywords: Multiple Dose Study in Overweight Healthy Subjects; body weight
MeSH Terms: conditions — Body Weight | interventions — PF-04620110

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04620110 (Experimental)
  Interventions: Drug: PF-04620110
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04620110 — Multiple oral doses of 5 mg of PF-04620110 will be given once daily for 2 weeks.
  Arms: PF-04620110
Drug: PF-04620110 — Multiple oral doses of 1.5 mg of PF-04620110 will be given twice daily for 2 weeks.
  Arms: PF-04620110
Drug: PF-04620110 — Multiple oral doses of 3 mg of PF-04620110 will be given once daily for 2 weeks.
  Arms: PF-04620110
Drug: PF-04620110 — Multiple oral doses of 2.5 mg of PF-04620110 will be given twice daily for 2 weeks.
  Arms: PF-04620110
Drug: Placebo — Multiple oral doses of placebo will be given once daily for 2 weeks.
  Arms: Placebo Comparator

SUMMARY:
PF-04620110 is a novel compound proposed for the treatment of Type 2 diabetes mellitus. The primary purpose of this trial is to evaluate the safety and tolerability, and pharmacodynamics, of multiple oral doses of PF-04620110.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years
* Body Mass Index (BMI) of 26.5 to 35.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To evaluate additional pharmacodynamic markers in response to multiple oral doses of PF-04620110. | Day 1 to Day 13
To evaluate secondary Pharmacodynamic Endpoints in response to a liquid meal test in response to multiple oral doses of PF-04620110. | Day 6 and Day 14

SECONDARY OUTCOMES:
To characterize the PK of PF-04620110 following multiple oral doses in otherwise healthy overweight and obese subjects. | Baseline to 2 weeks
To assess safety and tolerability of PF-04620110 will be assessed by physical examinations, adverse event monitoring, 12-lead ECGs, vital sign, and clinical safety laboratory measurements. | Baseline to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Investigational Site, Brussels, Belgium
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0961010&StudyName=A%20Multiple%20Dose%20Study%20Of%20PF-04620110%20In%20Healthy%20Overweight%20Or%20Obese%20Subjects